CLINICAL TRIAL: NCT04540094
Title: Feasibility of 5% Albumin Compared With Balanced Crystalloid, as Intravenous Fluid Resuscitation in Adult Patients With Sepsis, Presenting as an Emergency to Hospital: ABC Sepsis Trial
Brief Title: Feasibility of 5% Albumin Compared With Balanced Crystalloid, as Intravenous Fluid Resuscitation in Adult Patients With Sepsis, Presenting as an Emergency to Hospital
Acronym: ABC Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC20043
Record Dates: First submitted 2020-08-19; First posted 2020-09-07 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-08

CONDITIONS: Sepsis
Keywords: Sepsis; Emergency Care; Albumin; Crystalloid; Fluid; Resuscitation
MeSH Terms: conditions — Sepsis | interventions — Serum Albumin, Human

STUDY DESIGN:
Intervention Model Description: Open label two-arm, multicentre, pragmatic, parallel group randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5% Human Albumin Solution (Experimental): Participants allocated to the treatment arm will receive intravenous 5% Human Albumin Solution (HAS) administered as the sole intravenous fluid during the initial 6-hour resuscitation period. The clinician can deliver up to 10ml/kg in the first 3 hours using 250ml boluses of HAS based on clinical judgement, using clinical assessment supplemented by technology if that is their usual practice. This will be followed by repeat clinical assessment after each bolus (including vital signs; lactate testing). After 3 hours further HAS boluses up to 6 hours post-randomisation will be at clinical discretion and will be documented in the CRF. Patients in the albumin arm should not receive balanced crystalloid as a resuscitation fluid in the first 6 hours.
  Interventions: Drug: Human albumin
- Intravenous balanced crystalloid (Active Comparator): Participant allocated to the usual care arm will receive intravenous balanced crystalloid administered as the sole intravenous fluid during the initial 6 hour resuscitation period. The clinician can deliver up to 30ml/kg in the first 3 hours using 250ml boluses of balanced crystalloid based on clinical judgement, using clinical assessment supplemented by technology if that is their usual practice. This will be followed by repeat clinical assessment after each bolus (including vital signs; lactate testing). Thereafter, further crystalloid boluses up to 6 hours will be at the discretion of the clinical team and will be documented in the CRF. Patients in the balanced crystalloid arm should not receive albumin as a resuscitation fluid in the first 6 hours.
  Interventions: Drug: Balanced crystalloid solution

INTERVENTIONS:
Drug: Human albumin — Any preparation of 5% Human Albumin Solution which has marketing authorisation in the UK to be used for this indication and is stocked by local hospital pharmacies at the participating sites, may be prescribed in this study
  Arms: 5% Human Albumin Solution
Drug: Balanced crystalloid solution — Any preparation of intravenous "balanced" crystalloid which has marketing authorisation in the UK to be used for this indication and is stocked by local hospital pharmacies at the participating sites, may be prescribed in this study.
  Arms: Intravenous balanced crystalloid

SUMMARY:
The aim of this research study is to compare two different fluids (Human Albumin Solution (HAS) and Balanced Crystalloid that are given via a drip to patients with severe infection (sepsis). The investigators plan to see which fluid is better, and to see if they have a role in improving a patient's recovery time, reducing complications and the length of time they stay in hospital. This study plans to find out if there is evidence that one fluid is better overall to determine the need for a subsequent definitive trial.

DETAILED DESCRIPTION:
This trial will be an open label two-arm, multicentre, pragmatic, parallel group randomised trial of adult patients with community acquired sepsis recruited from the Emergency Department and Medical and Surgical Assessment Units across ~10 UK NHS Hospitals. The treatment phase will be the first 6 hours following randomisation. 30-day and 90-day follow up will be conducted using routine data only. The exception to this will be the first 50 patients enrolled in the study, Health Related Quality of Life (HRQoL) will be measured using the EQ-5D-5L at baseline, 7 days and at 180 days. At baseline, the participant or their relative will be asked to recall the quality of life 4 weeks prior to the index hospital admission. Questionnaires will be administered by direct patient completion or, postal or email survey with telephone follow up for non-responders after two mailings two weeks apart.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (18 years or older) who present to UK NHS hospitals with community acquired sepsis meeting all of the 4 criteria:

1. Clinically suspected or proven infection resulting in principal reason for acute illness;
2. NEWS score ≥5 (or NEWS2 if adopted in recruitment site);
3. Hospital presentation within last 12hrs; and
4. Clinician decision has been made that immediate (within 1 hour) intravenous fluid resuscitation is needed.

Exclusion Criteria:

1. >1 litre of intravenous crystalloid fluid or any intravenous HAS administered prior to eligibility assessment;
2. Requirement for immediate surgery (within one hour of eligibility assessment);
3. Chronic renal replacement therapy;
4. Known allergy/adverse reaction to HAS;
5. Balanced crystalloid or HAS not available;
6. Known adverse reaction to blood products;
7. Palliation/end of life care (explicit decision by patient/family/carers in conjunction with clinical team that any active treatment beyond symptomatic relief is not appropriate);
8. Religious beliefs precluding HAS administration;
9. Previous recruitment in the trial;
10. Known recent severe traumatic brain injury (within 3 months);
11. Patients with permanent incapacity;
12. Known recruitment in another CTIMP studies within the last 30 days where co-enrolment has not been agreed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Gray, Study Director — University of Edinburgh
Locations (15):
- United Kingdom (15):
  - Aberdeen Royal Infirmary, Aberdeen
  - Addenbrookes Hospital, Cambridge
  - Derby Teaching Hosptial NHS Foundation Trust, Derby
  - Royal Infirmary Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - St Johns, Livingston
  - St Georges Hospital, London
  - University College London Hospital, London
  - John Radcliffe Hospital, Oxford
  - Royal Alexandra Hospital, Paisley
  - Derriford Hospital Plymouth, Plymouth
  - Salford Royal NHS Foundation Trust, Salford
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
The intention is to share anonymised data with external collaborators and scientists one year after the primary publication has been published (anticipated Jun 2022).
Supporting Information: CSR, Analytic Code
Time Frame: From 2023
Access Criteria: Requests can be made by email to the Chief Investigator from 2023.

REFERENCES:
- [Derived] Gray AJ, Oatey K, Grahamslaw J, Irvine S, Cafferkey J, Kennel T, Norrie J, Walsh T, Lone N, Horner D, Appelboam A, Hall P, Skipworth RJE, Bell D, Rooney K, Shankar-Hari M, Corfield AR; Albumin, Balanced, and Crystalloid-Sepsis (ABC-Sepsis) Investigators. Albumin Versus Balanced Crystalloid for the Early Resuscitation of Sepsis: An Open Parallel-Group Randomized Feasibility Trial- The ABC-Sepsis Trial. Crit Care Med. 2024 Oct 1;52(10):1520-1532. doi: 10.1097/CCM.0000000000006348. Epub 2024 Jun 24. PMID 38912884

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (15) | 68 (18) | 69 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 70 | 149
  Male | 71 | 80 | 151
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Lactate [Mean (Standard Deviation); unit: mmol/l] | 3 (3) | 3 (2) | 3 (3)
National Early Warning Score (NEWS) Score [Mean (Standard Deviation); unit: units on a scale] — The National Early Warning Score (NEWS) was first introduced by the Royal College of Physicians in 2012 as a predictor of patient deterioration. It includes seven parameters (temperature, systolic blood pressure, respiratory rate, oxygen saturation, oxygen supply, heart rate, and level of consciousness). Each Parameter receives a score between 0-3 (+2 or 0 for supplemental oxygen Y/N) which correlates to severity and this is combined to create a total score. The score range is from 0 to 20. Patients are classified as a low score (NEWS 1-4), medium score (5-6) and high score (≥7).
  units on a scale | 8 (2.4) | 8.3 (2.7) | 8.1 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: We measured the recruitment rate to assess deliverability. We aimed to recruit 300 participants in approximately 1 year in a 1:1 ratio into each treatment arm.
Time Frame: Approx 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 150 | 150

2. Primary Outcome: 30-day Mortality
Description: Assessment of how many participants in each arm died after 30 days to determine the effect size between the treatment groups.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 147 | 149
Participants | 31 | 22

3. Secondary Outcome: Data Completeness of Primary Outcome
Description: Feasibility Outcome assessing the number of participants who provided data for clinical primary outcome (30 day mortality)
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 147 | 149

4. Secondary Outcome: Withdrawal From Study
Description: Feasibility Outcomes assessing the number of participants who withdraw from study intervention and/or data collection
Time Frame: Approx 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 3 | 1

5. Secondary Outcome: Number of Patients Who Receive Any Other Fluid Apart From Intervention or Control in First 6 Hrs After Recruitment
Description: Feasibility Outcome- number of patients who receive any other fluid apart from intervention or control in first 6 hrs after recruitment
Time Frame: 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 33 | 1

6. Secondary Outcome: Time to Start of In-hospital Intravenous Fluids
Description: Feasibility Outcome- Time to start of in-hospital intravenous fluids
Time Frame: From time of Randomisation until fluid first being administered measured up to 6 hours.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
minutes | 41 [17 to 76] | 36 [17 to 63]

7. Secondary Outcome: In-hospital Mortality
Description: Secondary Clinical Outcome
Time Frame: From time of Randomisation until time of hospital discharge or death, whichever is first measured up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 29 | 23

8. Secondary Outcome: 90-day Mortality
Description: Secondary Clinical Outcome
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 43 | 32

9. Secondary Outcome: Volume of Randomised Fluid Delivered in Each Arm in the First 6hrs
Description: Secondary Clinical Outcome- Volume of randomised fluid delivered in each arm in the first 6hrs
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
ml | 750 [500 to 1334] | 1250 [1000 to 2000]

10. Secondary Outcome: Length of Hospital Stay
Description: Secondary Clinical Outcome
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
days | 12.7 (15.9) | 13.9 (19.3)

11. Secondary Outcome: Proportion of Patients Admitted to Critical Care (HDU/ICU)
Description: Secondary Clinical Outcome- Proportion of patients admitted to critical care (HDU/ICU)
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 6 | 3

12. Secondary Outcome: Length of Stay in Critical Care (HDU/ICU)
Description: Secondary Clinical Outcome- Length of stay in critical care (HDU/ICU)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
days | 1.3 (5.9) | 1.5 (5.4)

13. Secondary Outcome: Number of Participants Needing Intravenous Vasopressors
Description: Secondary Clinical Outcome-number of participants needing intravenous vasopressors
Time Frame: From time of Randomisation until time of hospital discharge, measured up to 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 18 | 12

14. Secondary Outcome: Number of Participants Needing Renal Replacement
Description: Secondary Clinical Outcome- Number of participants needing renal replacement
Time Frame: From time of Randomisation until time of hospital discharge, measured up to 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 1 | 2

15. Secondary Outcome: Number of Participants Needing Invasive Ventilation
Description: Secondary Clinical Outcome- Number of participants needing invasive ventilation
Time Frame: From time of Randomisation until time of hospital discharge, measured up to 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 7 | 4

16. Secondary Outcome: Number of Patients Readmitted in First 90 Days After Discharge
Description: Secondary Clinical Outcome- Number of patients readmitted in first 90 days after discharge
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 20 | 21

17. Secondary Outcome: Number of Patients Developing Acute Kidney Injury (AKI)
Description: AKI Defined using National Institute for Health and Care Excellence (NICE) criteria:
  A diagnosis of AKI may be made if there is one of the following:
  A rise in serum creatinine of 26 micromol/L or greater within 48 hours. A 50% or greater rise in serum creatinine known or presumed to have occurred within the past 7 days.
  A fall in urine output to less than 0.5 mL/kg/hour for more than 6 hours.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 36 | 30

18. Secondary Outcome: Number of Patients Developing Pulmonary Oedema
Description: Safety Radiology diagnosis or requirement for rescue management (new diuretic use)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 22 | 11

19. Secondary Outcome: Number of Patients Developing Allergy or Anaphylaxis
Description: Requirement for rescue management (antihistamines, adrenaline, intravenous fluids, steroid)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
Participants | 0 | 1

20. Secondary Outcome: Health Related Quality of Life (EQ-5D-5L Questionnaire)
Description: Health Economic Outcomes are measured using the the 5-level EQ-5D version (EQ-5D-5L). The EQ-5D-5L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. A high score indicates a worse outcome. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. The digits for the five dimensions can be combined into a 5-digit number (profile) that describes the patient's health state. The EQ-5D profile can be converted to a single number between 0-1 called the EQ-5D value. These EQ-5D values to lie on between 0-1 to indicate health where 0 represents the minimum score (dead) and 1 is full health. Values less than 0 are possible for health states considered worse than dead.
Time Frame: baseline
Population: Health Related Quality of life questionnaires were applicable only to the first 50 participants who entered the study. As this is a self-reported questionnaire, participants may not be well enough to complete this at any given time-point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 19 | 26
score on a scale | 0.8 [0.2 to 0.9] | 0.5 [0.2 to 0.8]

21. Secondary Outcome: Secondary Care Costs
Description: Costs will be estimated by assigning national standard unit costs to inpatient stays (critical care and general ward level), readmissions and additional high costs activities observed in the study. Baseline (pre-admission) HQoL will be estimated using age/sex matched population reference data.
Time Frame: 30 days
Reporting Status: Not Posted

22. Secondary Outcome: Volume of Randomised Fluid Delivered in Each Arm in the First 24hrs
Description: Secondary Clinical Outcome-Volume of randomised fluid delivered in each arm in the first 24hrs
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 150 | 150
ml | 1012 (703) | 2209 (1461)

23. Secondary Outcome: Health Related Quality of Life (EQ-5D-5L Questionnaire)
Description: as for outcome 20
Time Frame: 7 Days
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 19 | 27
score on a scale | 0.4 [0.1 to 0.8] | 0.5 [0.2 to 0.7]

24. Secondary Outcome: Health Related Quality of Life (EQ-5D-5L Questionnaire)
Description: as for outcome 20
Time Frame: 180 Days
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
Number analyzed (Participants) | 20 | 28
units on a scale | 0.4 [0.1 to 0.8] | 0.5 [0.2 to 0.7]

ADVERSE EVENTS:
Time Frame: SAEs defined as outcome events were collected for 90 days. All other SAEs were collected for 7 days.
Description: All SAEs that meet the definition given in protocol section 11.1 and occur between consent and 7 days afterwards were recorded/reported to Sponsor. Outcome events are anticipated in this participant group were recorded for 90 days but exempt from reporting to the Sponsor:
  All-cause Death Death related to infection (including multi-organ failure) Critical care (HDU/ICU) admission Acute kidney injury Pulmonary oedema, Allergy or anaphylaxis
Arm/Group | 5% Human Albumin Solution | Intravenous Balanced Crystalloid
All-Cause Mortality (participants affected / at risk) | 43/150 | 32/150
Serious Adverse Events (participants affected / at risk) | 5/150 | 2/150
Other Adverse Events (participants affected / at risk) | 25/150 | 20/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5% Human Albumin Solution (N=150) | Intravenous Balanced Crystalloid (N=150)
General Disorders (General disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vascular Disorders (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5% Human Albumin Solution (N=150) | Intravenous Balanced Crystalloid (N=150)
Blood and Lymphatic (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Cardiac Disorders (Cardiac disorders) | 2 (2) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 0 (0)
General disorders and administration (General disorders) | 2 (2) | 2 (2)
Infections and infestations (Infections and infestations) | 0 (0) | 2 (2)
Investigations (Investigations) | 2 (2) | 5 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 2 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Full Health Economic Analysis was not possible to determine the difference in secondary care costs. It was determined that any comparative analysis of costs would be dominated by mortality difference between arms, with the inevitable lower costs and quality-adjusted life years (QALYs) associated with the higher mortality group, so full analysis of this data was not completed as it would not produce meaningful outcomes. All analyses outlined in the Statistical Analysis Plan were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04540094/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT04540094/SAP_001.pdf